CLINICAL TRIAL: NCT06633302
Title: Evaluating the Efficacy of a 26°C Indoor Temperature for Limiting Thermal and Cardiovascular Strain in Older Adults During a Simulated Multi-day Heat Event
Brief Title: Physiological Strain in Older Adults During a Simulated Heat Wave
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Professor, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HEPRU-2024-08-A
Record Dates: First submitted 2024-10-04; First posted 2024-10-09 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Heat Stress; Physiological Stress
Keywords: Heat wave; Indoor overheating; Indoor temperatures; Thermoregulation; Heat strain; Elderly; Heat vulnerability; Cardiovascular strain; Sleep; Hyperthermia; Fatigue
MeSH Terms: conditions — Heat Stress Disorders; Hyperthermia; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure to indoor temperature limits daylong (Experimental): Participants exposed to three consecutive days (3 days, 2 nights) in an indoor environment maintained at either 26°C at all times (condition A, recommended upper indoor temperature limits during an extreme heat event).
  Interventions: Other: Simulated multi-day heatwave exposure
- Exposure to indoor temperature limits nighttime only (Experimental): Participants exposed to three consecutive days (3 days, 2 nights) to indoor overheating during the daytime (34°C, temperatures experienced in homes without air-conditioning) (9:00 to 19:00) with nighttime (19:00 to 9:00) indoor temperatures reduced to the recommended limit of 26°C.
  Interventions: Other: Simulated multi-day heatwave exposure

INTERVENTIONS:
Other: Simulated multi-day heatwave exposure — Older adults exposed to a multi-day simulated heat wave exposure

SUMMARY:
A recent report showed that maintaining indoor temperature at or below 26°C safeguards older, heat vulnerable adults against potentially dangerous increases in thermal and cardiovascular strain during an extreme heat event (PMID: 38329752). However, this proposed limit does not consider the potential cumulative effect of successive days of heat exposure, which could lead to a progressive deterioration in thermoregulatory and cardiovascular function and necessitate adjustments to upper indoor temperature limits. Further, thermal comfort and quality of sleep may be negatively impacted when bedroom temperatures exceed 24°C (PMID: 3090680). On this basis, some health agencies have recommended that bedroom temperatures at night should not exceed 26°C unless ceiling fans are available (PMID: 3090680). Currently, however, it is unknown whether indoor overheating impairs sleep quality and physiological strain on a subsequent day in older adults and, if so, whether maintaining indoor temperature at 26°C is sufficient to prevent these adverse health impacts.

With rising global temperatures and more extreme heat events, energy management strategies to limit the strain on the power grid during the daytime are now increasingly commonplace. Thus, understanding the benefits of maintaining indoor temperature at the recommend upper limits of 26°C during the nighttime only on surrogate physiological indicators of health is an important step in understanding how to optimize protection for heat-vulnerable older adults when power outages occur.

The investigators will assess the efficacy of proposed indoor temperature limits (i.e., 26°C) in mitigating increases in core temperature and cardiovascular strain over three consecutive days (3 days, 2 nights) in older adults (60-85 years) with (indoor temperatures maintained at the recommend 26°C at all times throughout the three days) and without (daytime temperature fixed at 34°C (temperature experienced in homes without air-conditioning during an extreme heat event) with nighttime temperature at 26°C) access to daytime cooling. By quantifying the effect of daylong indoor overheating on surrogate physiological outcomes linked with heat-related mortality and morbidity in older adults, the investigators can determine if refinements in the recommended upper temperature threshold is required, including best practices when power outages may occur during an extreme heat event.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking.
* English or French speaking.
* Ability to provide informed consent.
* with or without a) chronic hypertension (elevated resting blood pressure; as defined by Heart and Stroke Canada and Hypertension Canada), b) type 2 diabetes as defined by Diabetes Canada, with at least 5 years having elapsed since time of diagnosis

Exclusion Criteria:

* Episode(s) of severe hypoglycemia (requiring the assistance of another person) within the previous year, or inability to sense hypoglycemia (hypoglycemia unawareness).
* Serious complications related to your diabetes (gastroparesis, renal disease, uncontrolled hypertension, severe autonomic neuropathy).
* Uncontrolled hypertension - BP >150 mmHg systolic or >95 mmHg diastolic in a sitting position.
* Restrictions in physical activity due to disease (e.g. intermittent claudication, renal impairment, active proliferative retinopathy, unstable cardiac or pulmonary disease, disabling stroke, severe arthritis, etc.).
* Use of or changes in medication judged by the patient or investigators to make participation in this study inadvisable.
* Cardiac abnormalities identified during screening

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Core temperature (Peak) during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Peak rectal temperature (15 min average) during exposure. Rectal temperature is measured continuously throughout the daytime period of the simulated heat wave.
Core temperature (AUC) during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Area under the curve of rectal temperature (in degree-hours)
Core temperature end of daytime exposure | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Rectal temperature measured at hour 10 of each daytime exposure to simulated heat wave (15-min average)
Heat rate peak during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Heart rate during each daytime exposure to simulated heat wave (15-min average)
Heat rate AUC during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Heart rate measured during each daytime exposure to simulated heat wave (15-min average)
Cardiac response to standing from supine (30:15 Ratio) during daytime | At the start (hour 0) and end of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Cardiac response to standing evaluated as the ratio between the highest R-wave to R-wave interval (lowest heart rate) measured at the 30th heart beat after standing from supine (+/- 5 beats) and the lowest R-wave to R-wave interval (highest heart rate) measured at the 15th heart beat after standing (+/- 5 beats). Cardiac response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest). Assessment is performed in the morning prior to and following daytime exposure.
Reaction time during daytime (cognitive function) | At the start (hour 0) and end of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of reaction time. Participants will be asked to initiate a movement of the device in response to a visual cue.
Impulse control during daytime (cognitive function) | At the start (hour 0) and end of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of impulse control. Participants will be asked to respond to both "go" and "no-go" visual cues. In response to the "go" cue, participants will initiate a movement of the device.
Memory recall during daytime (cognitive function) | At the start (hour 0) and end of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of memory recall. Participants complete both a delayed recall test and a working memory test.
Executive function during daytime (cognitive function) | At the start (hour 0) and end of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of executive function. Participants will complete the Cued Stroop test, in which they are presented a sequence of congruent, neutral and incongruent colour-word tasks.
CDC 4-Stage Balance Test during daytime (Postural stability) | At the start (hour 0) and end of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  To assess postural stability, participants hold a tablet to their chest, then auditory cues guide participants through four consecutive stances, feet side by side, instep of one foot touching the big toe of the other foot, tandem stand with one foot in front of the other, heel touching toe, and stand on one foot. The balance assessment will be evaluated based on movement detected by an accelerometer integrated into the hardware of the tablet device (Sway Medical Inc).
BTrackS Balance Assessment during daytime (Postural stability) | At the start (hour 0) and end of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  To assess postural stability, participants will be asked to stand on a BTracks force plate with their feet spread out to shoulder width, hand on their hips and eyes closed. The assessment will comprise of four trials (one practice trial) lasting 20 seconds in length and 20 seconds between trials. Center of pressure (COP) vector data along vertical (y) and horizontal (x) axes will be summed for the total path excursion length (cm) during each trial.
Systolic Response to Standing From Supine during daytime | At the start (hour 0) and end of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Systolic blood pressure response to standing evaluated as the difference in blood pressure measured between the standing and supine. Standing systolic blood pressure will be taken as the lowest value of those measured after 60 and 120 seconds of standing. Systolic response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest).
Systolic blood pressure during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Systolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures)
Diastolic blood pressure during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Diastolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures)
Rate pressure product during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Rate pressure product, an index of myocardial work and strain, calculated as systolic blood pressure x heart rate.
Heart rate variability: SDNN during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Standard deviation of normal-to-normal R-wave to R-wave intervals (SDNN) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the seated position. SDNN will be evaluated twice, during two paced breathing periods (separated by 4 min of seated rest).
Heart rate variability: RMSSD during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Root mean squared standard deviation of normal-to-normal R-wave to R-wave intervals (RMSSD) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the seated position. RMSSD will be evaluated twice, during two paced breathing periods (separated by 4 min of seated rest).
Fluid consumption during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Average hourly fluid consumption calculated by weighing participant water intake at the start and end of each hour of exposure (normalized to the exposure duration).
Fluid loss during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Fluid loss calculated as the change in body mass during each exposure presented as a percentage of baseline body mass (corrected for food consumption)
Change in plasma volume during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Change in plasma volume from baseline values calculated from duplicate measurements of hemoglobin and hematocrit at the start and end of each exposure using the technique by Dill and Costill
Thermal comfort scale during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Thermal comfort assessed via a visual analog scale ("How comfortable does your body temperature feel?") ranging from "extremely uncomfortable" to "extremely comfortable"(midpoint: neutral).
Thermal sensation scale during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Thermal sensation assessed via a visual analog scale ("How hot do you feel?") ranging from "extremely hot" to "neutral"(midpoint: hot)
Thirst sensation scale during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Thirst sensation scale assessed via a visual analog scale ("How thirsty are you?") ranging from "Very, very thirsty" to "Not thirsty at all" (midpoint: moderately thirsty).
Arousal scale during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Felt arousal scale assessed via a visual analog scale ("How worked up are you?") ranging from "high arousal" to "low arousal".
Orthostatic intolerance symptoms assessment during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Cumulative sum of scores on 6 questions asking participant to rank symptoms associated with orthostatic intolerance during the lying to standing tests. All symptoms scored on a scale from 0 (none) to 10 (worst possible) and include feelings of: (1) "dizziness, lightheadedness, feeling faint, or feeling like you might black out"; (2) "Problems with vision (blurring, seeing spots, tunnel vision, etc.)"; (3) "Weakness"; (4) "Fatigue"; (5) "Trouble concentrating"; and (6) "Head and neck discomfort".
Core temperature (Peak) during nighttime | End of nighttime exposure (hour 24 for Day 1 and Day 2 of the three day exposure; no nighttime exposure for Day 3) (daytime defined as period between 19:00 to 9:00)
  Peak rectal temperature (15 min average) during exposure. Rectal temperature is measured continuously throughout the daytime period of the simulated heat wave.
Core temperature (AUC) during nighttime | End of nighttime exposure (hour 24 for Day 1 and Day 2 of the three day exposure; no nighttime exposure for Day 3) (daytime defined as period between 19:00 to 9:00)
  Area under the curve of rectal temperature (in degree-hours)
Core temperature end of nighttime | End of nighttime exposure (hour 24 for Day 1 and Day 2 of the three day exposure; no nighttime exposure for Day 3) (daytime defined as period between 19:00 to 9:00)
  Rectal temperature measured at hour 10 of each daytime exposure to simulated heat wave (15-min average)
Heat rate peak during nighttime | End of nighttime exposure (hour 24 for Day 1 and Day 2 of the three day exposure; no nighttime exposure for Day 3) (daytime defined as period between 19:00 to 9:00)
  Heart rate during each daytime exposure to simulated heat wave (15-min average)
Heat rate AUC during nighttime | End of nighttime exposure (hour 24 for Day 1 and Day 2 of the three day exposure; no nighttime exposure for Day 3) (daytime defined as period between 19:00 to 9:00)
  Heart rate measured during each daytime exposure to simulated heat wave (15-min average)
Heart rate variability: SDNN during nighttime | End of nighttime exposure (hour 24 for Day 1 and Day 2 of the three day exposure; no nighttime exposure for Day 3) (daytime defined as period between 19:00 to 9:00)
  Standard deviation of normal-to-normal R-wave to R-wave intervals (SDNN) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the seated position. SDNN will be evaluated twice, during two paced breathing periods (separated by 4 min of seated rest).
Heart rate variability: RMSSD during nighttime | End of nighttime exposure (hour 24 for Day 1 and Day 2 of the three day exposure; no nighttime exposure for Day 3) (daytime defined as period between 19:00 to 9:00)
  Root mean squared standard deviation of normal-to-normal R-wave to R-wave intervals (RMSSD) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the seated position. RMSSD will be evaluated twice, during two paced breathing periods (separated by 4 min of seated rest).

SECONDARY OUTCOMES:
Muscle oxygen during battery of cardiovascular, postural and cognitive tests during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Participants will be attached with one probe placed on the left prefrontal cortex and one on the muscle belly of the vastus lateralis to measure tissue oxygenation using near-infrared spectroscopy (NIRS; Portalite, Artinis Medical, The Netherlands).
Profiles of Mood States (POMS) during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Potential changes in mood (7 subscales of mood: tension, anger, depression, fatigue, confusion, vigor and esteem-related affect). The POMS-40 is a validated, self-administered questionnaire that examines seven distinct aspects of mood state across two positive subscales (Esteem-Related Affect, and Vigor) and five negative subscales (Fatigue, Tension, Confusion, Anger, and Depression), which are described across 40 distinct adjectives. For each individual item, participants were asked to describe "how you feel right now" by responding using a 5-point Likert scale (0 = "Not at all", 1 = "A little", 2 = "Moderately", 3 = "Quite a lot", or 4 = "Extremely"). The values of items associated with a specific subscale (e.g., Fatigue) were summed to calculate its score.
Environmental Symptoms Questionnaire (ESQ) | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Self-reported environmental reactions and medical symptomatology associated with prolonged heat exposure. The ESQ-IV is a validated 68-item, self-administered questionnaire that has been used successfully in identifying symptomatology during exposure to a wide variety of environmental conditions, including heat exposure [24, 25]. Participants are asked to assess and described "how you have been feeling today" by responding to each item using a 6-point Likert scale (0 = "Not at all", 1 = "Slight", 2 = "Somewhat", 3 = "Moderate", 4 = "Quite a bit", or 5 = "Extreme"). Total Symptom Score was calculated from this data by taking the sum of the intensity ratings from all 68 individual items using reverse scores for the three positive items from the list ("I Felt Good", "I Felt Alert", and "I Felt Wide Awake").
Sleep quality and quantify assessment | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  The following questionnaires will be administered:
  Consensus Sleep Diary (CSD) to provide an overview of the sleep quantity and quality of the previous night.
  Richards-Campbell Sleep Questionnaire to evaluate the perception of sleep .
  Leeds Sleep evaluation questionnaire which is 10-item, subjective, questionnaire designed to assess changes in sleep quality over the course of the intervention.
Sleepiness during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  The following questionnaires will be administered to evaluate the participants sleepiness during the daytime exposure period:
  Karolinska sleepiness scale measures the subjective level of sleepiness at a particular time during the day.
  Stanford sleepiness scale consists of only one item, where participant must identify one of seven statements that best represents their level of perceived sleepiness

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada